CLINICAL TRIAL: NCT00500513
Title: Assessment of the Reliability of Implanted Fiducials for Tracking of Respiratory-Induced Tumor Motion
Brief Title: Tracking of Respiratory-Induced Tumor Motion Using Implanted Fiducials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0208
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Respiratory-Induced Tumor Motion; Tumor Motion; Pulmonary Function; Fiducial Marker
MeSH Terms: conditions — Lung Neoplasms | interventions — Fiducial Markers; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implanted Markers + CT + RT (Experimental)
  Interventions: Procedure: CT Scans; Procedure: Implanted markers; Radiation: Radiation Treatment (RT)

INTERVENTIONS:
Procedure: CT Scans — CT scan performed weekly to measure how much the tumor moves + additional pulmonary function measurements.
  Other Names: Computed Tomography; 4-D CT Scan
Procedure: Implanted markers — Implanted radio-opaque fiducial markers, diameter of 1.0 - 2.0 mm, inserted through a catheter at several chest locations using a flexible bronchoscope
Radiation: Radiation Treatment (RT) — Radiotherapy incorporating respiratory treatment delivery
  Other Names: RT; XRT

SUMMARY:
Objectives:

* To determine the safety of fiducial implantation.
* To determine the extent/rate of migration of radio-opaque fiducials placed in lung tumors and adjacent normal tissue.
* To compare real-time portal imaging-based fiducial tracking with measurement of three-dimensional motion by four-dimensional CT scanning to determine how many fiducials are needed to track a tumor.
* To determine if intra-fractional lung tumor motion changes during a course of treatment, and when during the treatment this occurs.
* To correlate the position of internal fiducials with the position of the external patient surface during respiration.
* To quantify the residual motion of the clinical target volume during radiotherapy gated using external fiducials.
* To verify the adequacy of the treatment portal margins in encompassing the residual motion of the clinical target volume.
* To determine if radio-opaque fiducial placement adjacent to the trachea (which does not move) can reduce daily setup inaccuracies, and so spare normal tissue.
* To determine the motion of hilar adenopathy (if any), and whether it correlates with motion of the primary tumor.

DETAILED DESCRIPTION:
If you are eligible to take part in this study, you will have pulmonary (lung) function testing. This testing will involve your breathing through a mouthpiece and measuring the amount of air you breathe. This will provide information on how well your lungs work, and how your chest wall moves when you breathe.

You will then begin the normal treatment planning process. A bean-bag "cast" will be made for you to lie in during planning and treatment. This is done to lower day-to-day changes in your position. A CT scan will be taken with you breathing quietly, and possibly several X-rays will be performed as well. You will be marked with magic marker, and possibly have several permanent tattoos placed to help with daily positioning. These procedures normally take 1-2 hours.

Small metal markers (up to 5) will then be placed near your tumor. A thin, flexible tube with a camera, called a bronchoscope, will be used to place these markers in your lungs. You will be given a sedative through one of your veins and a local anesthetic will be sprayed in your nose and mouth before introducing the bronchoscope. The bronchoscope is introduced through one of your nostrils and then passed into your windpipe and bronchial tubes. This will allow the doctor to examine your lungs and place the small metal markers. These markers will be used to track the tumor during treatment. In this way the radiation treatment can be given to the tumor even if it moves while you breathe.

You will also have studies to measure how much the tumor moves. This will be done with several additional CT scans, typically taken on a weekly basis. Additional pulmonary function measurements will be taken during the CT scans. These measurements will allow researchers to monitor the movement of your tumor when you breathe. These procedures will normally take between 1 and 2 hours.

You will be on this study for the duration of your radiation treatments. You will be followed up an for an additional 4 - 6 weeks to make sure there are no complications from the study.

THIS IS AN INVESTIGATIONAL STUDY. A total of up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be undergoing radiation treatment.
2. Planned course of radiation treatment must be greater than or equal to 6 weeks.
3. The patient is able to tolerate bronchoscopy: a. Able to maintain oxygen saturation >95% on room air nasal cannula supplementation <5L/min, b. Can tolerate supine position without respiratory difficulties, c. Has normal hemodynamic parameters, d. Has normal coagulation profile
4. The patient is a candidate for bronchogenic placement of seeds.
5. The patient has an identifiable tumor on a CT scan.
6. The patient has signed the consent form.

Exclusion Criteria:

1. The patient has had previous thoracic surgery (e.g., lobectomy, pneumonectomy, tumor excision). Biopsy, mediastinoscopy, mastectomy are not exclusions.
2. The patient has had previous radiation to the thorax.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-04; Primary Completion 2007-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing motion of one or more fiducials during the course of radiation therapy | Baseline, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Starkschall, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org